CLINICAL TRIAL: NCT01834547
Title: Phase I Study About Effects of Caffeine, Methylphenidate, Modafinil and Placebo on Cognitive Performance of Chess Players.
Brief Title: Cognitive Hyper-performance - Effects of Stimulating Substances in Chess-players
Acronym: CHESS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: K. Lieb (Other)
Responsible Party: Sponsor-Investigator, K. Lieb, Prof. Dr. med. K. Lieb, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1234
Record Dates: First submitted 2011-05-25; First posted 2013-04-18 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Cognitively Healthy Subjects Influenced by Psychoactive Drugs
Keywords: chess, cognition
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Methylphenidate (Experimental): Methylphenidate
  Interventions: Drug: Drugs use: methylphenidate
- modafinil (Experimental): modafinil
  Interventions: Drug: Drug use: modafinil
- caffeine (Experimental): caffeine
  Interventions: Drug: caffeine
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Drugs use: methylphenidate — 40 mg tablets
  Arms: Methylphenidate
Drug: Drug use: modafinil — 40 mg tablets
  Arms: modafinil
Drug: caffeine — 400 mg
  Arms: caffeine
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
Effects of caffeine, methylphenidate, modafinil and placebo on cognitive performance of chess players in chess games and neuropsychiatric standardized tests. We hypothesize that substances will change cognitive performance in chess players leading to changed results in chess games and neuropsychiatric tests.

ELIGIBILITY:
Inclusion Criteria:

* male
* 18-60 years old
* existence of ELO-number

Exclusion Criteria:

* physical diseases (e.g. diabetes mellitus, etc.) with necessity of using prescription drugs
* psychiatric diseases (e.g. psychosis, bipolar disorders, etc.) with necessity of using prescription drugs
* addiction of psychoactive substances
* smoker or quitter (< 5 years)
* use of more than 5 cups of coffee per day
* irregular day-night-rhythm (e.g. shift workers)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Chess games (win/ lose/ tie) | two years

SECONDARY OUTCOMES:
time period for decision of chess games | results of ches games
Cognitive performance measured with standardized neuropsychiatric tests (Tower of Hanoi, Trail-Making test, Stroop-Test, Psycho-Motor-Vigilance test, Wisconsin-Card-Sorting-Test, Balloon Analog Risk Task) | outcome of tests
measuring of risk taking behaviour, motivation, mood using standardized questionnaires | outcome of tests
adverse events | type of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Mainz, Germany